CLINICAL TRIAL: NCT03993353
Title: A Phase II Study of Tadalafil and Pembrolizumab in Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Tadalafil and Pembrolizumab in Recurrent or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Joseph Califano, Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190098
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma; Head and Neck Carcinoma; Head and Neck Cancer Stage III; Head and Neck Cancer Stage IV; Head and Neck Cancer Metastatic; Cancer; Cancer of Esophagus; Cancer, Metastatic; Cancer of Head and Neck; Cancer of Mouth; Cancer of Neck
Keywords: cancer; pembrolizumab; tadalafil; cialis; opdivo; immunotherapy; metastatic; carcinoma; pd-1; pde
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Neoplasms; Esophageal Neoplasms; Neoplasm Metastasis; Mouth Neoplasms; Carcinoma; Parkinson Disease 4, Autosomal Dominant Lewy Body; Pyridoxine-dependent epilepsy | interventions — pembrolizumab; Tadalafil

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tadalafil and Pembrolizumab (Experimental): Tadalafil for up to 12 months and pembrolizumab for up to 24 months.
  Interventions: Drug: Pembrolizumab; Drug: Tadalafil

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg intravenously every 3 weeks
  Other Names: Keytruda
Drug: Tadalafil — 10 mg by mouth daily
  Other Names: Cialis

SUMMARY:
This study will examine the combination of pembrolizumab and tadalafil for safety and efficacy in advanced head and neck cancer.

DETAILED DESCRIPTION:
Immune competent animal models of HNSCC demonstrate that combination PDE-5 inhibitor (tadalafil) and PD-1 inhibitor therapy is more effective than either therapy alone based on the concept of targeting multiple immune repressive abnormalities simultaneously (PD-1 checkpoint and myeloid suppressive pathways).

This trial will test the hypothesis that combination PD-1 inhibition and PDE-5 inhibition can be safely co-administered, and secondarily test the hypothesis that the combination of both therapies will be more effective than PD-1 inhibition alone in recurrent/metastatic HNSCC.

ELIGIBILITY:
Selected Inclusion Criteria:

* Patients (at least 18 years of age) must have recurrent or metastatic squamous cell carcinoma of the head and neck.
* Presence of measurable disease.
* Life expectancy of greater than 12 weeks
* Patients must have normal organ and marrow function

Selected Exclusion Criteria:

* Prior therapy with an PD-1 or PD-L1 inhibitor in the recurrent or metastatic setting
* Uncontrolled central nervous system metastases (stable metastases permitted)
* Active autoimmune disease
* Chemotherapy ≤28 days prior to first administration of study treatment and/or monoclonal antibody ≤8 weeks prior to first administration of study treatment.
* Prior daily use of tadalafil or other long-acting PDE5 inhibitors for one month or greater within 3 months of trial enrollment
* Current use of all other long-acting PDE5 inhibitors.
* Known severe hypersensitivity to tadalafil or any of the excipients of this product
* Current treatment with nitrates
* Current systemic treatment with a potent cytochrome P450 3A4 (CYP3A4) inhibitor such as ketoconazole or ritonavir.
* Current treatment with guanylate cyclase (GC) stimulators such as riociguat.
* History of hypotension and/or blindness and/or sensorineural hearing loss during prior treatment with tadalafil or other PDE-5 inhibitors
* History of known hereditary degenerative retinal disorders, including retinitis pigmentosa
* Prior history of non-arteritic anterior ischemic optic neuropathy
* Pregnant or breastfeeding; a negative pregnancy test is required within 14 days of randomization for all women of childbearing potential.
* History of stroke within prior 6 months.
* History of acute myocardial infarction within prior 3 months, uncontrolled angina, uncontrolled arrhythmia, or uncontrolled congestive heart failure
* Left ventricular outflow obstructions, such as aortic stenosis and idiopathic hypertrophic subaortic stenosis
* Angina requiring treatment with long-acting nitrates
* Angina requiring treatment with short-acting nitrates within 90 days of planned tadalafil administration
* Unstable angina within 90 days of visit 1 (Braunwald 1989)
* Positive cardiac stress test without documented evidence of subsequent, effective cardiac intervention
* History of any of the following coronary conditions within 90 days of planned tadalafil administration:

  * Myocardial Infarction
  * Coronary artery bypass graft surgery
  * Percutaneous coronary intervention (for example, angioplasty or stent placement)
  * Any evidence of heart disease (NYHA ≥ Class II as defined in Protocol Attachment LVHG.3) within 6 months of planned tadalafil administration
* Concurrent systemic immunosuppressant therapy (e.g., cyclosporine A, tacrolimus, etc., or chronic administration of >10 mg/day of prednisone or equivalent)
* Prior organ transplantation
* Known history of human immunodeficiency virus (HIV) or active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2022-04-16 (Actual); Study Completion 2024-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Califano, Principal Investigator — UCSD
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tadalafil and Pembrolizumab
Started | 7
Completed | 6
Not Completed | 1
Not completed — Screen Failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tadalafil and Pembrolizumab
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.67 (6.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 2
  Unknown or Not Reported | 0
Cancer Type [Count of Participants; unit: Participants]
  Hypopharynx | 1
  Larynx | 2
  Oral cavity | 2
  Oropharynx | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Dose Limiting Toxicity (DLT)
Description: Rate of dose limiting toxicity at least possibly attributable to study treatment
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Tadalafil and Pembrolizumab
Number analyzed (Participants) | 6
Participants | 1

2. Primary Outcome: Overall Survival (OS)
Description: Overall survival at 12 months post-enrollment
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tadalafil and Pembrolizumab
Number analyzed (Participants) | 6
Participants | 3

3. Secondary Outcome: Response Measured by RECIST 1.1
Description: Response measured by RECIST 1.1
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tadalafil and Pembrolizumab
Number analyzed (Participants) | 3
Participants | 1

4. Secondary Outcome: Progression Free Survival
Description: Progression free survival
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Tadalafil and Pembrolizumab
Number analyzed (Participants) | 3
months | 21.56 (22.98)

5. Secondary Outcome: Adverse Event Rates
Description: Adverse event rates
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Tadalafil and Pembrolizumab
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Tadalafil and Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 3/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil and Pembrolizumab (N=6)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil and Pembrolizumab (N=6)
Endocrine disorders (Endocrine disorders) | 1 (2)
Eye disorders (Eye disorders) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (9)
General disorders and administration site conditions (General disorders) | 4 (7)
Infections and infestations (Infections and infestations) | 3 (3)
Investigations (Investigations) | 1 (2)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3 (4)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (2)
Psychiatric disorders (Psychiatric disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 4 (5)
Vascular disorders (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT03993353/Prot_SAP_001.pdf